CLINICAL TRIAL: NCT06729801
Title: Intrarenal Pressure Monitoring Via Flexible and Navigable Suction Ureteral Access Sheath in Retrograde Intrarenal Surgery: A Pilot Clinical Study
Brief Title: Intrarenal Pressure Monitoring Via Flexible and Navigable Suction Ureteral Access Sheath in Retrograde Intrarenal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERE2024-003
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Kidney Stone
Keywords: RIRS; FANS
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRP-Monitoring FANS Group (Experimental): Patients in this group will undergo retrograde intrarenal surgery (RIRS) using the intrarenal pressure (IRP)-monitoring flexible and navigable suction ureteral access sheath (FANS). This novel device provides real-time IRP monitoring, enabling the surgeon to adjust intraoperative irrigation and suction settings to optimize stone retrieval efficiency while maintaining IRP within a safe range.
  Interventions: Device: IRP-Monitoring Flexible and Navigable Suction Ureteral Access Sheath (FANS)
- Conventional FANS Group (Active Comparator): Patients in this group will undergo RIRS using a conventional flexible and navigable suction ureteral access sheath (FANS) without intrarenal pressure (IRP) monitoring. The irrigation flow rate and suction pressure will be pre-set and adjusted based on standard clinical practices.
  Interventions: Device: Conventional FANS

INTERVENTIONS:
Device: IRP-Monitoring Flexible and Navigable Suction Ureteral Access Sheath (FANS) — The IRP-Monitoring Flexible and Navigable Suction Ureteral Access Sheath (FANS) is a novel device designed to enable real-time monitoring of intrarenal pressure (IRP) during retrograde intrarenal surgery (RIRS). It incorporates a pressure-sensing port connected to a gas conduit embedded in the sheath, which allows the surgeon to adjust irrigation flow and suction pressure based on real-time IRP readings, thereby optimizing stone retrieval efficiency while ensuring safety by maintaining a safe IRP range. The device improves surgical outcomes, particularly in complex cases involving larger renal stones, by reducing operative time and minimizing the risk of complications.
  Arms: IRP-Monitoring FANS Group
Device: Conventional FANS — The Conventional Flexible and Navigable Suction Ureteral Access Sheath (FANS) is a standard device used in retrograde intrarenal surgery (RIRS) for stone retrieval. Unlike the IRP-monitoring version, this device does not provide real-time monitoring of intrarenal pressure (IRP). Irrigation flow and suction pressure are pre-set and adjusted based on clinical protocols. It facilitates the removal of renal stones through a flexible and navigable design, but without the added capability of monitoring and adjusting IRP during the procedure.
  Arms: Conventional FANS Group

SUMMARY:
This study evaluates the use of a novel intrarenal pressure (IRP)-monitoring flexible and navigable suction ureteral access sheath (FANS) in retrograde intrarenal surgery (RIRS) for renal stones. The prospective clinical trial compares its efficacy and safety against conventional FANS in 100 patients. The primary outcomes include IRP monitoring accuracy, operative time, stone-free rate (SFR), and complication rates, with the aim of improving stone retrieval efficiency and procedural safety in RIRS. This trial seeks to validate the innovative device's role in expanding RIRS indications, especially for large renal stones.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-75 years old) diagnosed with renal stones (size ≤4 cm) and suitable for retrograde intrarenal surgery (RIRS).
2. Willing to provide informed consent.
3. No significant renal, cardiac, or systemic diseases that may interfere with the surgical procedure or the study.
4. Preoperative intravenous pyelography (IVP) showing no significant ureteral stricture.

Exclusion Criteria:

1. Patients with active urinary tract infections (UTIs) or fever at the time of surgery.
2. Pregnancy or breastfeeding women.
3. Patients with a history of severe renal disease (e.g., chronic kidney disease stage 3 or higher).
4. History of prior ureteral or renal surgery that may affect the anatomy.
5. Patients with uncontrolled comorbidities such as uncontrolled diabetes, hypertension, or cardiovascular disease.
6. Patients who are unwilling or unable to comply with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Operative Time | Measured during the surgical procedure, from the start of the surgery to the end of the procedure (estimated duration: 30-60 minutes per patient).
  The primary outcome will be the total operative time, measured from the insertion of the endoscope into the urethra to the completion of stent placement. This outcome will assess the efficiency of stone retrieval when using either the IRP-monitoring FANS or the conventional FANS.

SECONDARY OUTCOMES:
Stone-Free Rate (SFR) | 24-48 hours post-surgery, based on CT scan results.
  The stone-free rate (SFR) will be measured postoperatively through non-contrast CT imaging. The SFR will assess the effectiveness of stone retrieval and the success of the procedure.
Postoperative Complications | Evaluated within 30 days post-surgery.
  The rate of postoperative complications, including fever, infection, bleeding, or ureteral injury, will be recorded. This will help compare the safety profile of both FANS devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Guohua Zeng, Guangzhou, Guangdong, China